CLINICAL TRIAL: NCT04904809
Title: Perclose Multi-Access DUS Study: Assess the Safety and Performance of the Perclose ProGlide™ Suture-Mediated Closure (SMC) System and the Perclose™ ProStyle™ Suture-Mediated Closure and Repair (SMCR) System in Managing Multiple Venous Access Sites (Evaluation by DUS)
Brief Title: Perclose Multi-Access Duplex Ultrasound (DUS) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10410
Record Dates: First submitted 2021-05-18; First posted 2021-05-27 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Arrhythmia
Keywords: ABT-CIP-10410; Ablation; DUS; Femoral DUS
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All Registered Patients (Experimental): All registered patients will have multiple access sites in a single vein closed utilizing the Perclose ProGlide SMC System and/or Perclose ProStyle SMCR System.
  Interventions: Device: Perclose ProGlide SMC System and/or Perclose ProStyle SMCR System

INTERVENTIONS:
Device: Perclose ProGlide SMC System and/or Perclose ProStyle SMCR System — The Perclose ProGlide SMC and Perclose ProStyle SMCR in this study will be used for multiple access site closures in a single vein in the ablation procedure.
  Other Names: Perclose ProStyle SMCR System

SUMMARY:
The aim of this prospective, single-arm, United States (US) multi-center, descriptive clinical study is to evaluate the safety of multiple access site closure in a single vein with the SMC System by scheduled DUS at discharge and at 30 days (if vascular complications observed at discharge) in asymptomatic or non-visible subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Subject is planned to have an ablation procedure that requires multiple sheaths insertion in a single femoral vein
* All the access sites are planned to be treated with Perclose SMC
* Written informed consent is obtained prior to the procedure

Exclusion Criteria:

* Visible vascular thrombus (angiographic or ultrasound) in the ipsilateral leg prior to the ablation procedure
* Prior ipsilateral deep vein thrombosis within 6 months
* International Normalization Ratio >3.5 for patients on warfarin
* Subject who is not able to ambulate pre-procedure
* Women who are pregnant (based on site standard pre-procedure pregnancy test)
* Has active symptoms and/or a positive test result of COVID-19 or other rapidly spreading novel infectious agent within the prior 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjaya K Gupta, MD, Principal Investigator — St. Luke's Hospital; Soroosh Kiani, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - St. Luke's Hospital, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 36 subjects will be registered at 2 US investigational sites. All subjects must have femoral duplex ultrasound (DUS) at discharge and at a 30-dayfollow-up visit (if any access site-related vascular complications(either symptomatic/visible or asymptomatic/nonvisible), nerve injury, or infection at discharge, by either the investigator or the core laboratory).
Groups:
- All Registered Patients: All registered patients will have multiple access sites in a single vein closed utilizing the Perclose ProGlide suture-mediated closure (SMC) System and/or Perclose ProStyle suture-mediated closure and repair (SMCR) System.
  Perclose ProGlide SMC System and/or Perclose ProStyle SMCR System: The Perclose ProGlide SMC and Perclose ProStyle SMCR in this study will be used for multiple access site closures in a single vein in the ablation procedure.
Period: Overall Study
Arm/Group | All Registered Patients
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study enrolled a total of 36 subjects at 2 investigational sites.
Arm/Group | All Registered Patients
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1
Arrhythmia [Count of Participants; unit: Participants]
  Paroxysmal AF | 17
  Persistent AF | 11
  Atrial Flutter | 6
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Major Vascular Complications by DUS Detection at Discharge
Description: Vascular complications detected by scheduled DUS at discharge in subjects with asymptomatic/non-visible complications. Major complications are defined as those which require surgical, interventional, or pre-specified repair and/or hospitalization.
Time Frame: Within 24 hours of procedure.
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Registered Patients
Number analyzed (Participants) | 32
Participants
  Femoral Vein Stenosis (> 50%) Development at the Puncture | 0
  Deep Vein Thrombosis in the Target Limb | 0
  Hematoma | 0
  Pseudoaneurysm | 0
  Requiring Surgical or Percutaneous Repair | 0
  Requiring Thrombin Injection, Fibrin Adhesive Injection, or Ultrasound-guided Compression | 0
  Arteriovenous (AV) Fistula | 0
  Venous Tear | 0
  Venous Perforation | 0
  Arterial Tear | 0
  Arterial Perforation | 0
  Other Vascular Complication | 0
  Arterial Stenosis | 0
  Arterial Dissection | 0
  Mobile Perclose Common Femoral Vein | 0

2. Primary Outcome: Number of Subjects With Minor Vascular Complications by DUS Detection at Discharge
Description: Vascular complications detected by scheduled DUS at discharge in subjects with asymptomatic/non-visible complications. All complications other than Major complications are considered to be minor complications.
Time Frame: Within 24 hours of procedure.
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Registered Patients
Number analyzed (Participants) | 32
Participants
  Femoral Vein Stenosis (> 50%) Development at the Puncture Site related to Closure Techniqu | 0
  Deep Vein Thrombosis in the Target Limb | 3
  Hematoma | 1
  Pseudoaneurysm | 0
  Arteriovenous (AV) Fistula | 0
  Venous Tear | 0
  Venous Perforation | 0
  Arterial Tear | 0
  Arterial Perforation | 0
  Other Vascular Complication | 1
  Arterial Stenosis | 0
  Arterial Dissection | 0
  Mobile Perclose Common Femoral Vein | 1

ADVERSE EVENTS:
Time Frame: 30 days
Description: The data reported/presented under Outcome Measure 2 is a list of "vascular complications", whereas data reported under "Other (Not Including Serious) Adverse Events" section is a list of adverse events. In this study, there was 1 subject with deep vein thrombosis (DVT) that was identified by the site, reported as adverse event, and adjudicated by the CEC. In addition, there were 2 subjects that had DVT identified by the DUS core lab but not identified by the site.
Arm/Group | All Registered Patients
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 1/36
Other Adverse Events (participants affected / at risk) | 5/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Registered Patients (N=36)
Oesophagitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Registered Patients (N=36)
Vascular Access (Injury, poisoning and procedural complications) | 1
Site Haemorrhage (Injury, poisoning and procedural complications) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Venous Haemorrhage (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT04904809/Prot_SAP_001.pdf